CLINICAL TRIAL: NCT07309809
Title: Portrait Mobile Monitoring Solution V2.0 External Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SA-000173
Record Dates: First submitted 2025-12-03; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Monitoring
Keywords: Continuous Monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous Monitoring with Portrait Mobile (Experimental): Subjects will be monitored with the Portrait Mobile Monitoring Solution for up to 72 hours
  Interventions: Device: Continuous Monitoring

INTERVENTIONS:
Device: Continuous Monitoring — Subjects will have vital signs continuously monitored for up to 72 hours with the study device

SUMMARY:
The purpose of this study is to collect and assess feedback from the users regarding the functionality and performance of the Portrait Mobile Monitoring Solution V2.0. In addition, this study aims to collect raw parameter data from the investigational devices for use in current and future Portrait Mobile development, including engineering purposes as deemed appropriate by the Sponsor.

DETAILED DESCRIPTION:
Subjects will be enrolled from a general hospital ward to receive continuous monitoring for up to 72 hours by the Portrait Mobile Monitoring Solution V2.0. After the completion of that monitoring, both the clinician and the subject will complete a feedback survey about their experience with the device. The surveys along with raw data from the device will be collected from each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is age 18 years or older (≥18 years).
2. Participant must have the ability to understand and provide written informed consent.
3. Are being cared for in a hospital unit and are expected to remain in the unit for the duration of the study procedure.
4. Participant must be willing and able to comply with study procedures and duration.

Exclusion Criteria:

1. Known to be pregnant and/or breast feeding.
2. Diagnosed with infection requiring isolation.
3. Are immunocompromised.
4. Have previously participated in this study (no subject may participate more than once).
5. Subjects with Implantable Minute Ventilation Rate Responsive Pacemakers should be excluded from respiration rate monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Collection of user feedback surveys from Clinicians | Up to 72 hours
  Number of clinician feedback surveys collected at the end of each shift for clinicians overseeing care of subjects receiving continuous vital signs monitoring.
Collection of Subject Survey | up to 72 hours
  Number of subject surveys collected from study participants at the end of their continuous monitoring

SECONDARY OUTCOMES:
Collection of raw parameter data from Portrait Mobile Device | up to 72 hours
  Collection of electronic waveforms and device logs from the investigational device for the entire monitoring period for each subject.

CONTACTS AND LOCATIONS:
Locations (1):
- West Middlesex University Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No